CLINICAL TRIAL: NCT01695681
Title: Screen-detected Coeliac Disease. Prevalence and Impact on Gastrointestinal Symptoms and Quality of Life
Brief Title: Screen-detected Coeliac Disease, a Population Based Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Norwegian Coeliac Society (Unknown); The Gastrointestinal Research Foundation, University Hospital of NorthNorway (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/1943 (REK)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Celiac Disease
Keywords: Quality of life; Celiac Disease/diet therapy; Celiac Disease/diagnosis; Prospective Studies
MeSH Terms: conditions — Celiac Disease; Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary instruction (Other): Gluten-free diet
  Interventions: Other: Gluten-free diet

INTERVENTIONS:
Other: Gluten-free diet — Dietary advice by clinical dietitian

SUMMARY:
The purpose of this study is to determine the prevalence of previously undiagnosed coeliac disease based on a health survey from Tromsø, Norway. Moreover, the health impact of undiagnosed coeliac disease will be examined.

DETAILED DESCRIPTION:
Few population-based studies have examined the prevalence of coeliac disease and the impact of undiagnosed coeliac disease on health. Moreover, the number of people with undiagnosed coeliac disease is much higher than the number who know their diagnosis.

The purpose of this study is to determine the prevalence of coeliac disease and the impact of undiagnosed coeliac disease on health.

In a health survey of the population of Tromsø Norway, serological markers of coeliac disease (transglutaminase 2, TG2 and deamidated gliadin antibody test) have been analyzed. Individuals with increased level of one of these markers, will be invited for upper endoscopy with small bowel biopsy examination to confirm the diagnosis of coeliac disease. All persons with screen detected coeliac disease, will be advised to start a gluten free diet.

Health status and Quality of Life will be examined by means of the Gastrointestinal Symptoms Rating Scale (GSRS) and the Psychological General Well-Being Index (PGWBI) respectively.

1. At baseline GSRS and PGWBI will be analyzed in persons with screen detected and biopsy verified coeliac disease and compared with a group of healthy control persons from the health-survey cohort.
2. In a prospective study of the persons with screen detected coeliac disease, health status (GSRS) and Quality of Life will be compared before and after one year on a gluten free diet.

ELIGIBILITY:
Inclusion Criteria:

* Increased level of serological markers (Transglutaminase 2 or Deamidated Gliadin) and biopsy verified coeliac disease

Exclusion Criteria:

* Previously diagnosed coeliac disease

Ages: 30 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-04-15 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms: Gastrointestinal symptoms rating scale (GSRS) | 7 days
  The Gastrointestinal symptoms rating scale (GSRS) is a disease-specific instrument with 15 items combined into five major domains: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation.
  The scale assesses symptom severity using a seven-grade Likert scale, ranging from 1 (no discomfort at all) to 7 (very severe discomfort). A lower score indicates less symptoms.
  GSRS is obtained at first visit and at follow-up (>one year) to evaluate change in one of the five domain scores or total score (primary outcome)

SECONDARY OUTCOMES:
Quality of life score: Psychological General Well-Being Index (PGWBI) | 7 days
  The Psychological General Well-Being Index (PGWBI) is a generic instrument with 22 items combined into six major domains: Anxiety, Depressed Mode, Positive well-being, Self-control, General Health and Vitality
  The scale assesses symptom severity from 0 to 5. Higher score indicates a better psychological well being.
  PGWB is obtained at first visit and at follow-up (>one year) to evaluate change in one of the six domains or total score (secondary outcome)
Self-reported change in abdominal complaints | One year
  Retrospective assessment at follow-up: The participants with diagnosed celiac disease were asked about abdominal complaints after the change to a gluten-free diet. The question was answered on a 7-grade Likert scale from "very much worse" to "very much better"
Self-reported change in energy | One year
  Retrospective assessment at follow-up: The participants with diagnosed celiac disease were asked about energy/feeling-fit after the change to a gluten-free diet. The question was answered on a 7-grade Likert scale from "very much worse" to "very much better"

CONTACTS AND LOCATIONS:
Overall Officials: Jan- M Kvamme, MD PhD, Principal Investigator — University of Tromso; Trond Halstensen, MD PhD, Study Chair — University of Oslo
Locations (1):
- University hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Kvamme JM, Sorbye S, Florholmen J, Halstensen TS. Population-based screening for celiac disease reveals that the majority of patients are undiagnosed and improve on a gluten-free diet. Sci Rep. 2022 Jul 25;12(1):12647. doi: 10.1038/s41598-022-16705-2. PMID 35879335